CLINICAL TRIAL: NCT05442580
Title: Phase 1 Study of Lintivirally Transduced T Cells Engineered to Contain Anti-CD38 Linked to TCRζ and 4-1BB Signaling Domains in Subjects With Acute Myeloid Leukemia and Multiple Myeloma
Brief Title: CART-38 in Adult AML and MM Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administrative decision
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC# 19422
Record Dates: First submitted 2022-06-28; First posted 2022-07-05 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia (AML); Multiple Myeloma (MM)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Multiple Myeloma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Intervention Model Description: Three dose levels of CART-38 cells will be evaluated using a 3+3 dose escalation design in two parallel disease cohorts as follows:
  * Cohort A: Relapsed/Refractory Acute Myeloid Leukemia (AML)
  * Cohort B: Multiple Myeloma (MM)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort A Dose Level 1: Relapsed/Refractory Acute Myeloid Leukemia (AML) (Experimental): Cohort A Dose Level 1: Adult patients ages ≥ 18 with acute myeloid leukemia (AML) who have not achieved remission after at least two lines of prior therapy will receive a single fixed dose of 3x10(6) CART 38 Cells via intravenous infusion on Day 0, following lymphodepleting chemotherapy with cyclophosphamide or fludarabine based on physician discretion.
  Interventions: Drug: 3x10(6) CART-38 cellls; Drug: Cyclophosphamide; Drug: Fludarabine
- Cohort A Dose Level -1 :Relapsed/Refractory Acute Myeloid Leukemia (AML) (Experimental): Cohort A Dose Level -1: Adult patients ages ≥ 18 with acute myeloid leukemia (AML) will receive a single fixed dose of 7x10(5) CART 38 Cells via intravenous infusion on Day 0, following lymphodepleting chemotherapy with cyclophosphamide or fludarabine based on physician discretion.
  Interventions: Drug: 7x10(5) CART-38 cells; Drug: Cyclophosphamide; Drug: Fludarabine
- Cohort A Dose Level 2 :Relapsed/Refractory Acute Myeloid Leukemia (AML) (Experimental): Cohort A Dose Level 2: Adult patients ages ≥ 18 with acute myeloid leukemia (AML) will receive a single fixed dose of 7x10(6) CART 38 Cells via intravenous infusion on Day 0, following lymphodepleting chemotherapy with cyclophosphamide or fludarabine based on physician discretion.
  Interventions: Drug: 7x10(6) CART-38 cells; Drug: Cyclophosphamide; Drug: Fludarabine
- Cohort A Dose Level 3 :Relapsed/Refractory Acute Myeloid Leukemia (AML) (Experimental): Cohort A Dose Level 3: Adult patients ages ≥ 18 with acute myeloid leukemia (AML) will receive a single fixed dose of 3x10(7) CART 38 Cells via intravenous infusion on Day 0, following lymphodepleting chemotherapy with cyclophosphamide or fludarabine based on physician discretion.
  Interventions: Drug: 3x10(7) CART-38 cells; Drug: Cyclophosphamide; Drug: Fludarabine
- Cohort B Dose Level 1: Multiple Myeloma (MM) (Experimental): Cohort B Dose Level 1 - Adult patients ages ≥ 18 with Multiple Myeloma (MM) who have not achieved remission after at least two lines of prior therapy will receive a single fixed dose of 3x10(6) CART 38 Cells via intravenous infusion on Day 0, following lymphodepleting chemotherapy with cyclophosphamide or fludarabine based on physician discretion.
  Interventions: Drug: 3x10(6) CART-38 cellls; Drug: Cyclophosphamide; Drug: Fludarabine
- Cohort B Dose Level -1: Multiple Myeloma (MM) (Experimental): Cohort B Dose Level -1 - Adult patients ages ≥ 18 with Multiple Myeloma (MM) who have not achieved remission after at least two lines of prior therapy will receive a single fixed dose of 7x10(5) CART 38 Cells via intravenous infusion on Day 0, following lymphodepleting chemotherapy with cyclophosphamide or fludarabine based on physician discretion.
  Interventions: Drug: 7x10(5) CART-38 cells; Drug: Cyclophosphamide; Drug: Fludarabine
- Cohort B Dose Level 2: Multiple Myeloma (MM) (Experimental): Cohort B Dose Level 2 - Adult patients ages ≥ 18 with Multiple Myeloma (MM) who have not achieved remission after at least two lines of prior therapy will receive a single fixed dose of 7x10(6) CART 38 Cells via intravenous infusion on Day 0, following lymphodepleting chemotherapy with cyclophosphamide or fludarabine based on physician discretion.
  Interventions: Drug: 7x10(6) CART-38 cells; Drug: Cyclophosphamide; Drug: Fludarabine
- Cohort B Dose Level 3: Multiple Myeloma (MM) (Experimental): Cohort B Dose Level 3 - Adult patients ages ≥ 18 with Multiple Myeloma (MM) who have not achieved remission after at least two lines of prior therapy will receive a single fixed dose of 3x10(7) CART 38 Cells via intravenous infusion on Day 0, following lymphodepleting chemotherapy with cyclophosphamide or fludarabine based on physician discretion.
  Interventions: Drug: 3x10(7) CART-38 cells; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: 3x10(6) CART-38 cellls — 3x10(6) CART-38 cells via intravenous infusion
  Arms: Cohort A Dose Level 1: Relapsed/Refractory Acute Myeloid Leukemia (AML); Cohort B Dose Level 1: Multiple Myeloma (MM)
Drug: 7x10(5) CART-38 cells — 7x10(5) CART-38 cells via intravenous infusion
  Arms: Cohort A Dose Level -1 :Relapsed/Refractory Acute Myeloid Leukemia (AML); Cohort B Dose Level -1: Multiple Myeloma (MM)
Drug: 7x10(6) CART-38 cells — 7x10(6) CART-38 cells via intravenous infusion
  Arms: Cohort A Dose Level 2 :Relapsed/Refractory Acute Myeloid Leukemia (AML); Cohort B Dose Level 2: Multiple Myeloma (MM)
Drug: 3x10(7) CART-38 cells — 3x10(7) CART-38 cells via intravenous infusion
  Arms: Cohort A Dose Level 3 :Relapsed/Refractory Acute Myeloid Leukemia (AML); Cohort B Dose Level 3: Multiple Myeloma (MM)
Drug: Cyclophosphamide — Lymphodepleting chemotherapy administered at physician discretion
Drug: Fludarabine — Lymphodepleting chemotherapy administered at physician discretion

SUMMARY:
This is an open-label Phase 1 study to estimate the safety and manufacturing feasibility of lentivirally transduced T cells expressing anti-CD38 chimeric antigen receptors expressing tandem TCRζ and 4-1BB (TCRζ /4-1BB) costimulatory domains in patients with Acute Myeloid Leukemia and Multiple Myeloma. This CAR T cell product will be referred to as "CART-38 cells".

DETAILED DESCRIPTION:
This is an open-label Phase 1 study to estimate the safety and manufacturing feasibility of lentivirally transduced T cells expressing anti-CD38 chimeric antigen receptors expressing tandem TCRζ and 4-1BB (TCRζ /4-1BB) costimulatory domains in patients with Acute Myeloid Leukemia and Multiple Myeloma. This CAR T cell product will be referred to as "CART-38 cells".

Three dose levels of CART-38 cells will be evaluated using a 3+3 dose escalation design in two parallel disease cohorts as follows:

* Cohort A: Relapsed/Refractory Acute Myeloid Leukemia (AML)
* Cohort B: Multiple Myeloma (MM)

Enrollment in Cohorts A and B may occur in parallel, however subject infusions must be staggered as follows:

* Inter-Cohort Stagger: The first three subjects in the study, irrespective of cohort assignment, must be staggered by a minimum of 28 days.
* Intra-Cohort Stagger: In order to allow for appropriate monitoring/assessment of toxicities, the 1st and 2nd subject infusions at every dose level within each individual disease cohort must be staggered by at least 28 days. If there are no emergent safety concerns identified in the first subject infused, subsequent subject infusions within that disease cohort/dose level do not need to be staggered and may be infused sequentially (e.g. 2nd and 3rd subject infusions may occur in parallel). Formal DLT evaluations will be performed after the 3rd subject in each disease cohort/dose level reaches the Day 28 safety follow-up visit, and will allow for a formal decision regarding dose level progression, expansion, or de-escalation. Formal DLT evaluations will be determined by the Clinical PI and Sponsor Medical Director.

Cohort-specific DLT assessments will be performed after the 3rd evaluable subject at each dose level completes their Day 28 Safety Follow-up Visit. Generally, each cohort/dose level will be evaluated as follows. Please refer to Section 3.1 of the study protocol for complete details:

* If 0 DLTs are observed in the first 3 DLT evaluable subjects at an assigned dose level, the disease cohort will advance to the next dose level. If 0 DLTs are observed in the first 3 DLT evaluable subjects at the highest dose level (Dose Level 3), the disease cohort will add an additional 3 DLT evaluable subjects at this dose level to further evaluate safety.
* If 1 DLT is observed in the first 3 DLT evaluable subjects at an assigned dose level, the disease cohort will enroll an additional 3 evaluable subjects at this dose level to further evaluate safety. If 0 DLTs are observed in the second 3 evaluable subjects at this dose level (or a total of 1 DLT/6 evaluable subjects), the disease cohort will advance to the next dose level.
* If 2 DLTs are observed at an assigned dose level at any time, enrollment into that disease cohort will be stopped and the dose level for that cohort will be de-escalated to the previous dose level. If fewer than 6 DLT evaluable subjects were infused at the previous dose level, up to 6 total evaluable subjects will be infused to establish the maximum tolerated dose (MTD).
* The MTD is defined as the dose at which 0 or 1 DLT occurs in 6 DLT evaluable subjects.

DLT evaluable subjects are those who receive CART-38 cells as per their assigned dose level and either a) complete the DLT evaluation period per protocol, or b) experience a DLT that requires premature study discontinuation during the DLT evaluation period. Subjects that do not qualify as DLT evaluable will be replaced at the same dose level.

Retreatment:

Subjects who have demonstrated clinical benefit after their initial CART-38 infusion may also be eligible to receive retreatment with CART-38 cells at the physician-investigator's discretion. The CART-38 retreatment dose administered must not exceed a CART-38 dose that has been fully explored at previous dose levels and established as safe. Therefore, retreatment will remain closed until the safety of the CART-38 cells has been fully established within Dose Level 1 for that Cohort, and DSMB and FDA approval to open retreatment has been received.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients age ≥ 18 years.
2. Patients must have one of the following diagnoses:

   a. Cohort A: Acute Myeloid Leukemia (AML) which meets one of the following criteria: i. Patients with second or greater relapse defined as flow cytometric confirmation of myeloid leukemia of at least 0.1% after second documented complete remission; OR ii. Patients with detectable disease post-allogeneic transplant with flow cytometric confirmation (MRD) of myeloid leukemia of at least 0.1%; OR iii. Patients with refractory disease defined as persistent bone marrow involvement with >5% blasts after two courses of induction chemotherapy for patients at initial presentation or >5% bone marrow blasts after one course of re-induction chemotherapy for patients who have relapsed after previously achieving a complete remission; OR iv. Patients with relapsed disease (defined as >5% bone marrow blasts after one course of standard chemotherapy) after previously achieving a complete remission. Note: Two cycles of combination therapy with a hypomethylating agent and venetoclax is considered one course of standard AML chemotherapy for the purpose of this criteria.

   b. Cohort B: Relapsed/refractory multiple myeloma (MM) according to IMWG 2016 criteria which meets the following conditions: i. Relapsed/refractory disease after receiving ≥ 3 lines of therapy, to ensure the patient has been exposed to ≥ 1 IMiD®, ≥ 1 proteasome inhibitor, and daratumumab; where refractory MM is defined as the achievement of less than a partial response (< PR after ≥ 2 cycles) and relapsed MM requires patients be ≤ 12 months from the last dose of their prior treatment regimen to confirmation of relapse) AND ii. Patients must also have measurable disease as defined by one of the following:

1. Serum M-protein ≥ 0.5 g/dL; 2. Urine M-protein ≥ 200 mg/24 hours; 3. Serum free light chain (FLC) assay; involved FLC level ≥ 100 mg/L provided the serum FLC ratio is abnormal; 4. ≥ 30% clonal plasma cells in the bone marrow aspirate or biopsy sample; 5. Measurable plasmacytomas > 2 cm in cross sectional diameter.

3. AML only: Documentation of CD38 Expression on leukemic blasts by flow or by immunohistochemistry (IHC). Results must be confirmed after last documented relapse and after any CD38-directed therapy (if applicable).

4. Confirmed availability of cells for a rescue transplant as a therapeutic back-up option as follows:

1. Cohort A (AML): Patients must have a suitable stem cell donor available who may donate cells in the event the subject needs to undergo an allogeneic HSCT. Donor may be matched or mismatched and must be found to be suitable according to the institution's standard criteria; donors must be fully cleared to proceed as the donor.
2. Cohort B (MM): Previously harvested autologous stem cells > 2x106/kg CD34+ cells.

   5. Adequate organ function defined as:

a. Creatinine ≤ 2.5 mg/dl or Creatinine Clearance > 30ml/min b. ALT/AST ≤ 5x upper limit of normal range c. Direct bilirubin ≤ 2.0 mg/dl, unless the subject has Gilbert's syndrome (≤3.0 mg/dl) d. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygen > 92% on room air e. Left Ventricle Ejection Fraction (LVEF) ≥ 40% confirmed by ECHO/MUGA

6. ECOG Performance Status that is either 0 or 1. 7. Signed informed consent form 8. Subjects of reproductive potential must agree to use acceptable birth control methods.

Exclusion Criteria:

1. Evidence of active hepatitis B or active hepatitis C. The following would not qualify as an active infection, thus would not exclude the subject from participating:

   1. Positive HBV serology with undetectable viral load and ongoing antiviral prophylaxis for potential HBV reactivation.
   2. Positive HCV serology with quantitative PCR for plasma HCV RNA below the lower limit of detection, with or without concurrent antiviral HCV treatment
2. Any active, uncontrolled infection
3. Severe, active co-morbidity that in the opinion of the physician-investigator would preclude participation in this study.
4. Class III/IV cardiovascular disability according to the New York Heart Association Classification
5. Patients with known somatic JAK2 V617F mutation by PCR or next generation sequencing.
6. Patients < 3 months from prior autologous transplant or < 6 months from prior allo ASCT .
7. Active acute or chronic GVHD requiring systemic therapy.
8. Dependence on systemic steroids or immunosuppressant medications.
9. Active CNS disease. patients with a history of CNS involvement that was successfully treated are eligible. Additional CNS testing such as a lumbar puncture and/or brain imaging is only required for eligibility if a subject is experiencing signs/symptoms of CNS involvement.
10. Pregnant or nursing (lactating) women.
11. Patients with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system, and unrelated to their cancer or previous cancer treatment.
12. Active autoimmune disease requiring systemic immunosuppressive treatment equivalent to ≥ 10mg daily equivalent of prednisone. Patients with autoimmune neurologic diseases (such as MS) will be excluded.
13. Known history of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-02-09 (Actual); Study Completion 2025-02-09 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with treatment related adverse events using NCI Common Terminology Criteria for Adverse Events (CTCAE) V5.0 | 15 years
Number of subjects with dose-limiting toxicities | 12 months
Determination of maximum tolerated dose assessed by collection of adverse events as graded by CTCAE. | 12 months

SECONDARY OUTCOMES:
Proportion of subjects who enroll on the study who receive study treatment | 12 months
Proportion of product release failures | 12 months
Frequency of manufacturing failures as determined by production of study treatment that meets protocol defined targeted dose | 12 months
Overall Response Rate (ORR) | 12 months
Overall Survival (OS) | 15 years
Progression-free Survival (PFS) | 15 years
Best Overall Response (BOR) | 15 years
Duration of Response (DOR) | 15 years
Need for HSCT or alloHSCT | 15 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States